CLINICAL TRIAL: NCT06861062
Title: Effects of Vitamin D3 and Yeast Beta-Glucan Supplementation on Glycemic Control and Cardiovascular Disease Risk in Patients With Type 2 Diabetes: A Randomized Double-Blind Controlled Trial
Brief Title: Effects of Vitamin D3 and Yeast Beta-Glucan Supplementation on Glycemic Control and Cardiovascular Disease Risk in Patients With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, An Pan, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VD, Yeast β-Glucan in Diabetes
Record Dates: First submitted 2025-02-23; First posted 2025-03-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Vitamin D; yeast β-glucan; Diabetes Mellitus, Type 2; Cardiovascular Disease; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D + yeast β-glucan (Active Comparator)
  Interventions: Drug: Vitamin D3; Dietary Supplement: yeast β-glucan
- Vitamin D + yeast β-glucan placebo (Active Comparator)
  Interventions: Drug: Vitamin D3; Dietary Supplement: yeast β-glucan placebo
- yeast β-glucan +Vitamin D placebo (Active Comparator)
  Interventions: Dietary Supplement: yeast β-glucan; Dietary Supplement: Vitamin D placebo
- Vitamin D placebo + yeast β-glucan placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin D placebo; Dietary Supplement: yeast β-glucan placebo

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3(cholecalciferol),1600 IU per day.
  Other Names: cholecalciferol
  Arms: Vitamin D + yeast β-glucan; Vitamin D + yeast β-glucan placebo
Dietary Supplement: yeast β-glucan — yeast β-glucan, 600mg per day.
  Arms: Vitamin D + yeast β-glucan; yeast β-glucan +Vitamin D placebo
Dietary Supplement: Vitamin D placebo — Vitamin D placebo
  Arms: Vitamin D placebo + yeast β-glucan placebo; yeast β-glucan +Vitamin D placebo
Dietary Supplement: yeast β-glucan placebo — yeast β-glucan placebo
  Arms: Vitamin D + yeast β-glucan placebo; Vitamin D placebo + yeast β-glucan placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled trial involving 2,500 individuals aged 40-79 with type 2 diabetes (T2D). The trial includes a 2-year intervention period followed by a 3-year post-intervention follow-up. The primary objective is to investigate (a) the effect of daily supplementation with vitamin D3 (1600 IU) or yeast β-glucan (600 mg) on glycemic control in patients with T2D and (b) whether daily supplementation with vitamin D3 (1600 IU) or yeast β-glucan (600 mg) reduces the predicted 10 year risk of atherosclerotic cardiovascular disease (ASCVD) in patients with T2D. The secondary objectives include evaluating the effects of vitamin D3 or yeast β-glucan supplementation on cardiometabolic risk factors, inflammatory markers, and liver and kidney function indicators, and assessing whether such supplementation reduces the risk of cardiovascular disease, microvascular complications and mortality over the 3-year post-intervention period.

DETAILED DESCRIPTION:
The goal of this randomized, double-blind, placebo-controlled trial, with a 2×2 factorial design in individuals with type 2 diabetes (T2D), is to investigate (a) the effect of daily dietary supplementation with vitamin D3 (1600 IU) or yeast β-glucan (600 mg) on glycemic control in patients with T2D and (b) whether vitamin D3 (1600 IU) or yeast β-glucan (600 mg) supplementation reduces the predicted 10 year risk of atherosclerotic cardiovascular disease (ASCVD) in patients with T2D. Approximately 2,500 subjects aged 40-79 with T2D will be included in this study. Eligible participants will be randomly assigned to one of four groups: (1) daily vitamin D3 (1600 IU) and yeast β-glucan (600 mg); (2) daily vitamin D3 (1600 IU) and placebo for yeast β-glucan; (3) daily placebo for vitamin D3 and yeast β-glucan (600 mg); or (4) daily placebo for vitamin D3 and placebo for yeast β-glucan. At baseline, questionnaires will be administered to collect data on sociodemographic factors, lifestyle habits, health status, cognitive function, and medical conditions, et al. Participants will also undergo physical measurements, and blood, urine, and feces samples will be collected at study centers. The study includes a 2-year intervention period followed by a 3-year post-intervention follow-up. Participants in all groups will take four capsules daily for 2 years: two capsules containing either vitamin D or its placebo and two capsules containing either yeast β-glucan or its placebo. During the 2-year intervention period, questionnaires, physical measurements, and sample collection will be conducted at 6, 12, and 24 months. This trial will also evaluate the effects of supplementation on cardiometabolic risk factors, inflammatory markers, and liver and kidney function indicators, and assess whether it reduces the risk of cardiovascular disease, microvascular complications, and mortality over the 3-year post-intervention period, providing scientific evidence for the health effects of vitamin D or yeast β-glucan in the T2D population.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus diagnosed by a physician based on the diagnostic criteria outlined in the Guideline for the Prevention and Treatment of Diabetes Mellitus in China (2024 Edition);
2. Men or women aged 40-79 years;
3. Convenient access to the study centers and permanent residence in the vicinity for the next five years;
4. Voluntary participation and signed written informed consent.

Exclusion Criteria:

1. History of clinical cardiovascular disease (including myocardial infarction, treatment or hospitalization for heart failure, stroke, and coronary revascularization) within the past 6 months;
2. History of severe diabetic microvascular complications (diabetic nephropathy with an estimated glomerular filtration rate (eGFR) < 30 mL/(min·1.73m²), proliferative diabetic retinopathy, confirmed diabetic peripheral neuropathy with abnormal nerve conduction studies or small fiber neuropathy testing);
3. History of cancer, excluding non-melanoma skin cancer or cancers with a favorable prognosis;
4. History of kidney stones, hypercalcemia, or hyperparathyroidism;
5. History of severe liver disease, severe kidney disease, severe gastrointestinal disease, severe infectious diseases, severe sarcoidosis or other granulomatous diseases, severe mental illness, or any other condition considered unsuitable for participation judged by the clinic team;
6. Laboratory evaluation:

   * Blood calcium levels greater than or equal to the normal range for the clinical site's laboratory;
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels higher than 3 times the normal range for the clinical site's laboratory;
   * eGFR < 30 mL/(min·1.73m²);
7. Individuals currently taking vitamin D supplements (>400 IU/day), calcium supplements (>600 mg/day), yeast β-glucan supplements (>250 mg/day), or those with a history of allergy or intolerance to vitamin D or prebiotic products;
8. Participation in other clinical trials within the past 3 months;
9. Planning to become pregnant within the next five years, or currently pregnant or breastfeeding.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | 24 months
  Change in HbA1c from baseline to the 24-month visit
Cardiovascular disease risk | 24 months
  Change in 10-year ASCVD risk score from baseline to the 24-month visit, assessed using China-PAR score, with a score range of 0-100%, where a higher score means a higher ASCVD risk

SECONDARY OUTCOMES:
Blood 25(OH)D | 24 months
  Change in blood 25(OH)D concentrations from baseline to the 24-month visit
Major cardiovascular events | 60 months
  Time to the first occurrence of any of the following: myocardial infarction, hospitalized or treated heart failure, stroke, revascularization of coronary arteries, or cardiovascular deaths
Microvascular disease | 60 months
  Time to the first occurrence of any of the following: nephropathy, retinopathy, or neuropathy
All-cause mortality | 60 months
  Deaths from any causes
Change in fasting plasma glucose | 24 months
  Change in fasting plasma glucose from baseline to the 24-month visit. The value is reported in millimole per liter (mmol/L).
Change in fasting C-peptide | 24 months
  Change in fasting C-peptide from baseline to the 24-month visit. The value is reported in nanogram per milliliter (ng/mL).
Change in insulin | 24 months
  Change in insulin from baseline to the 24-month visit. The value is reported in microunit per milliliter (μU/mL).
Change in HOMA-IR | 24 months
  Change in HOMA-IR from baseline to the 24-month visit. HOMA-IR = [Fasting Serum Insulin (μU/mL) × Fasting Plasma Glucose (mmol/L)] / 22.5. Lower values indicate better insulin sensitivity.
Change in Lipid profile | 24 months
  Change in total cholesterol, triglycerides, LDL-cholesterol, and HDL-cholesterol from baseline to the 24-month visit. These values are reported in millimole per liter (mmol/L).
Change in Liver function markers | 24 months
  Change in alanine aminotransferase (ALT), aspartate aminotransferase (AST), a nd gamma-glutamyl transferase (GGT) from baseline to the 24-month visit. These values are reported in units per liter (U/L).
Change in serum creatinine | 24 months
  Change in serum creatinine from baseline to the 24-month visit. The value is reported in micromole per liter (μmol/L).
Change in cystatin C | 24 months
  Change in cystatin C from baseline to the 24-month visit. The value is reported in milligram per liter (mg/L).
Change in eGFR | 24 months
  Change in estimated glomerular filtration rate (eGFR) from baseline to the 24-month visit. The CKD-EPI (2009) method to estimate eGFR value. The value is reported in milliliter per minute per 1.73 square meters (mL/min/1.73 m²).
Change in blood calcium | 24 months
  Change in blood calcium from baseline to the 24-month visit. The value is reported in millimole per liter (mmol/L).
Change in body weight | 24 months
  Change in body weight from baseline to the 24-month visit. The value is reported in kilogram (kg).
Change in BMI | 24 months
  Change in body mass index (BMI) from baseline to the 24-month visit. BMI = Body Weight (kg) / [Height (m)]^2. The value is reported in kilogram per square meter (kg/m^2).
Change in waist circumference | 24 months
  Change in waist circumference from baseline to the 24-month visit. The value is reported in centimeter (cm).
Change in waist-to-hip ratio | 24 months
  Change in waist-to-hip ratio from baseline to the 24-month visit. Waist-to-hip ratio = Waist Circumference (cm) / Hip Circumference (cm). Higher values indicate greater central adiposity.
Change in blood pressure | 24 months
  Change in systolic and diastolic blood pressure from baseline to the 24-month visit. The values are reported in millimeters of mercury (mmHg).
Change in grip strength | 24 months
  Change in grip strength from baseline to the 24-month visit, assessed using a handgrip dynamometer. The value is reported in kilogram (kg).
Change in FRAIL scale | 24 months
  FRAIL scale comprises five domains: fatigue, resistance, ambulation, illnesses, and weight loss. Each item is scored as 0 or 1, yielding a total score ranging from 0 to 5, with higher scores indicating greater frailty. Based on the total score, patients were categorized as robust (0 points), pre-frail (1-2 points), or frail (3-5 points).
Change in C-reactive protein | 24 months
  Change in C-reactive protein (CRP) from baseline to the 24-month visit. The value is reported in milligram per liter (mg/L).
Change in procalcitonin | 24 months
  Change in procalcitonin from baseline to the 24-month visit. The value is reported in nanogram per milliliter (ng/mL).
Change in interleukin-6 | 24 months
  Change in interleukin-6 (IL-6) from baseline to the 24-month visit. The value is reported in picogram per milliliter (pg/mL).
Bone mineral density | 24 months
  Change in bone mineral density from baseline to the 24-month visit, including but not limited to Speed of Sound (SOS), T-score, and Z-score. SOS is reported in meters per second （m/s). T-score and Z-score have no dimensional units.
Change in baPWV | 24 months
  Change in brachial-Ankle Pulse Wave Velocity (baPWV) from baseline to the 24-month visit. The value is reported in centimeters per second (cm/s).
Change in ABI | 24 months
  Change in Ankle-Brachial Index (ABI) from baseline to the 24-month visit. ABI=Systolic blood pressure of the ankle (mmHg) / Higher values of bilateral arm systolic pressure (mmHg).
Change in LSM | 24 months
  Change in stiffness measurement (LSM) from baseline to the 24-month visit, assessed by transient elastography (FibroTouch). The value is reported in kilopascal (kPa).
Change in UAP | 24 months
  Change in Ultrasound Attenuation Parameter (UAP) from baseline to the 24-month visit, assessed by transient elastography (FibroTouch). The value is reported in Decibel per Megahertz per Centimeter (dB/MHz/cm).

OTHER OUTCOMES:
Other events | 60 months
  Incidence of other cardiovascular diseases (not listed above), cancer, infectious diseases and falls
Change in Health-related quality of life | 24 months
  Change in health-related quality of life from baseline to the 24-month visit, assessed using EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire, with a score range of 0-100, where a higher score means higher health-related quality of life
Change in Cognitive function (MoCA) | 24 months
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA). The MoCA is a one-page 30-point test. Scores range from 0 to 30, with a score of 26 or above considered normal. The change in score from baseline to 24 months will be calculated.
Change in Cognitive function (MMSE) | 24 months
  Cognitive function will be assessed using the Mini-Mental State Examination (MMSE). The MMSE is a 30-point questionnaire. Scores range from 0 to 30, with different cut-off points for normal cognition based on education level: >17 for illiterate, >20 for individuals with ≤6 years of education, and >24 for individuals with >6 years of education. The change in score from baseline to 24 months will be calculated.
Change in depressive mood score | 24 months
  Change in depressive symptom severity from baseline to the 24-month visit, measured by the Patient Health Questionnaire-9 (PHQ-9) score, with a score range of 0-27, where a higher score means more severe depressive symptoms.
Change in anxiety score | 24 months
  Change in anxiety symptom severity from baseline to the 24-month visit, measured by the Generalized Anxiety Disorder-7 (GAD-7) score, with a score range of 0-21, where a higher score means more severe anxiety symptoms and clinical cut point for anxiety disorder was 10 points.
Change in Sleep quality | 24 months
  Change in sleep quality from baseline to the 24-month visit, assessed using the Pittsburgh Sleep Quality Index (PSQI), with a score range of 0-21, where a higher score means worse sleep quality.
Change in BF% | 24 months
  Change in body fat percentage (BF%) from baseline to the 24-month visit.
Change in fat mass | 24 months
  Change in fat mass from baseline to the 24-month visit. The value is reported in kilogram (kg).
Change in fat-free mass | 24 months
  Change in fat-free mass from baseline to the 24-month visit. The value is reported in kilogram (kg).
Concentration of blood metabolites | 24 months
  Blood metabolites, including, but not limited to, fatty acids and lipoprotein particles, quantified by liquid chromatography-tandem mass spectrometry (LC-MS/MS), are reported in mmol/L.
Metagenomic analysis of the gut microbiota | 24 months
  The diversity of the gut microbiota will be assessed by high-quality whole-metagenomic sequencing
DNA methylation level | 24 months
  The relative change in DNA methylation level quantified by pyrosequencing, reported as percentage methylation at specific CpG sites

CONTACTS AND LOCATIONS:
Overall Officials: An Pan, PHD, Principal Investigator — School of Public Health, Tongji Medical College, Huazhong University of Science and Technology
Locations (5):
- China (5):
  - Guangxi Medical College, Nanning, Guangxi
  - Kailuan General Hospital, Tangshan, Hebei
  - Sinopharm Dongfeng General Hospital, Shiyan, Hubei
  - Huazhong University of Science and Technology, Wuhan, Hubei
  - Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) sharing will need to be approved by the Institutional Review Board (IRB) and the study investigators with individual specific project request.